CLINICAL TRIAL: NCT01906489
Title: Phase 2b Randomized, Double-Blind, Placebo-Controlled Study to Assess the Pharmacodynamic Response, Safety, and Tolerability to 20 Weeks of Oral Dosing of AKB-6548 in Participants With Anemia Secondary to Chronic Kidney Disease (CKD), GFR Categories G3a-G5 (Stages 3, 4, AND 5) (Pre-Dialysis)
Brief Title: 20-Week Repeat Oral Dose Study of AKB-6548 in Participants With Chronic Kidney Disease and Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0007
Record Dates: First submitted 2013-07-20; First posted 2013-07-24 (Estimated); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-06

CONDITIONS: Anemia; Chronic Kidney Disease
Keywords: anemia; chronic kidney disease; CKD; chronic renal insufficiency; renal impairment; erythropoietin; kidney; oral anemia treatment; hemoglobin; hypoxia-inducible factor; HIF; hypoxia-inducible factor prolyl-hydroxylase inhibitor; HIF-PHI; efficacy; safety; pharmacokinetics
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Renal Insufficiency | interventions — vadadustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AKB-6548 (Experimental)
  Interventions: Drug: AKB-6548
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AKB-6548 — Oral dose administered once daily for 20 weeks. Dose adjustment based on hemoglobin level as defined in the protocol.
  Arms: AKB-6548
Drug: Placebo — Oral Placebo administered once daily for 20 weeks. Dose adjustment based on hemoglobin level as defined in the protocol.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the hemoglobin response (efficacy), safety, and tolerability of orally administered AKB-6548 in participants with Chronic Kidney Disease (pre-dialysis) with anemia with dosing for 20 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 to 82 years of age, inclusive
* Chronic Kidney Disease with a GFR category of G3a-G5 and not yet on dialysis
* eGFR ≥ 10 and ≤ 65 mL/minute/1.73 m2
* Anemia secondary to CKD with an ESA status and a Screening HGB as per protocol
* Iron replete with ferritin and TSAT levels as defined per protocol

Key Exclusion Criteria:

* BMI > 44.0 kg/m2
* Red blood cell transfusion within 11 weeks prior to the Screening visit
* Androgen therapy within the previous 21 days prior to the Screening visit
* Intravenous iron within the past 4 weeks prior to the Screening visit
* AST or ALT >1.8x ULN, alkaline phosphatase >2x ULN, or total bilirubin >1.5x ULN
* Screening ECG with QTc > 500 msec
* Uncontrolled hypertension
* Class III or IV congestive heart failure
* Myocardial infarction, acute coronary syndrome, or stroke within 6 months prior to the Screening visit

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2013-07-23 (Actual); Primary Completion 2014-09-03 (Actual); Study Completion 2014-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Akebia Therapeutics Inc.
Locations (47):
- United States (47):
  - Glendale, Arizona
  - Tucson, Arizona
  - Azusa, California
  - Chula Vista, California
  - Downey, California
  - El Centro, California
  - La Mesa, California
  - Long Beach, California
  - Riverside, California
  - Sacramento, California
  - San Diego, California
  - Arvada, Colorado
  - Westminster, Colorado
  - Lauderdale Lakes, Florida
  - Port Charlotte, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Macon, Georgia
  - Meridian, Idaho
  - Evergreen Park, Illinois
  - Lafayette, Louisiana
  - Shreveport, Louisiana
  - Detroit, Michigan
  - Lansing, Michigan
  - Petoskey, Michigan
  - Pontiac, Michigan
  - Farmington, Missouri
  - Kansas City, Missouri
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Flushing, New York
  - Mineola, New York
  - New Rochelle, New York
  - Rosedale, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Rocky Mount, North Carolina
  - Wilmington, North Carolina
  - Cincinnati, Ohio
  - Columbia, South Carolina
  - Knoxville, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Edinburg, Texas
  - Houston, Texas
  - San Antonio, Texas
  - St. George, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Pergola PE, Spinowitz BS, Hartman CS, Maroni BJ, Haase VH. Vadadustat, a novel oral HIF stabilizer, provides effective anemia treatment in nondialysis-dependent chronic kidney disease. Kidney Int. 2016 Nov;90(5):1115-1122. doi: 10.1016/j.kint.2016.07.019. Epub 2016 Sep 17. PMID 27650732

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 210 participants entered the study and 209 were randomized in a 2:1 ratio to receive Vadadustat or Placebo. However, 1 participant received Placebo in error.
Groups:
- Vadadustat: Participants received Vadadustat 450 milligrams (mg), as 3 tablets once daily (QD) for 20 consecutive weeks. The dose of study medication was increased to a maximum of 600 mg/day or decreased to 150 mg/day based on Hgb response. Participants received an iron supplement to maintain ferritin levels.
- Placebo: Participants received matching Placebo, as 3 tablets once daily (QD) for 20 consecutive weeks. Placebo was provided as white to off-white, oval film-coated tablets for oral administration. Participants received an iron supplement to maintain ferritin levels.
Period: Overall Study
Arm/Group | Vadadustat | Placebo
Started | 138 | 72
Completed | 112 | 63
Not Completed | 26 | 9
Not completed — Adverse Event | 10 | 3
Not completed — Worsening of CKD | 6 | 4
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Worsening of Anemia | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Non- Compliance | 1 | 0
Not completed — Sponsor Decision | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vadadustat | Placebo | Total
Number analyzed (Participants) | 138 | 72 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (9.97) | 65.9 (12.33) | 66.4 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 34 | 115
  Male | 57 | 38 | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 49 | 19 | 68
  White | 83 | 49 | 132
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Successful Hemoglobin Response
Description: Hemoglobin (Hgb) response was defined as participants with mean Hgb ≥11.0 grams per deciliter (g/dL) (average of Weeks 19 and 20) or increase in Hgb by ≥ 1.2 g/dL (average of Weeks 19 and 20) over pre-dose average (average of the two Hgb values obtained prior to dosing) without receiving Erythropoiesis-Stimulating Agents (ESA) or transfusion.
Time Frame: Weeks 19 and 20
Population: Per Protocol (PP) Population: participants in modified intent-to-treat (MITT) Population who had completed the study and had efficacy data through Week 20, had a study medication compliance of ≥ 80%, and did not have any protocol deviations. Only participants with available data were analyzed.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo: Participants were randomized to receive matching Placebo administered as 3 tablets once daily (QD) for 20 consecutive weeks. Placebo was provided as white to off-white, oval film-coated tablets for oral administration. Participants received an iron supplement to maintain ferritin levels.
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 102 | 58
Percentage of participants | 54.9 | 10.3
Statistical Analysis 1: Comparison: Vadadustat vs Placebo; Test type: Superiority; p = 0.0001, Fisher Exact; Odds Ratio (OR) = 11.4739, 95% CI 2-sided [3.3505 to 39.2931]

2. Secondary Outcome: Percentage of Participants With Hemoglobin Value ≥13.0 g/dL at Any Time During the Study
Description: Participants who have experienced an excursion in Hgb to ≥13.0 g/dL at any time during the study were considered as "failures". Data was presented for failures.
Time Frame: Up to 20 Weeks
Population: Modified Intent-to-Treat (MITT) Population: all randomized participants who received at least one dose of study medication and had a Baseline (either screening or Baseline for both Hgb and RBC count) and at least one post-Baseline measurement for both Hgb and RBC. Only participants with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 136 | 72
Percentage of participants | 59.6 | 88.9
Statistical Analysis 1: Comparison: Vadadustat vs Placebo; Test type: Other; p < 0.0001, Fisher Exact

3. Secondary Outcome: Percentage of Participants Achieving a Successful Hemoglobin Response, Determined Solely Based on the Hemoglobin Value
Description: Hgb response was defined as participants with mean Hgb ≥11.0 g/dL (average of Weeks 19 and 20) or increase in Hgb by ≥ 1.2 g/dL (average of Weeks 19 and 20) over pre-dose average (average of the two Hgb values obtained prior to dosing). Analysis of this secondary outcome measure is a reanalysis of the primary outcome measure whereby the response was determined solely by the Hgb value and receiving rescue therapy did not make the participant a failure.
Time Frame: Weeks 19 and 20
Population: MITT Population. Only participants with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 136 | 72
Percentage of participants | 44.9 | 13.9
Statistical Analysis 1: Comparison: Vadadustat vs Placebo; Test type: Other; p < 0.0001, Fisher Exact

4. Secondary Outcome: Percentage of Participants Achieving a Successful Hemoglobin Response in ESA Treatment naïve Group
Description: Hgb response was defined as participants with mean Hgb ≥11.0 g/dL (average of Weeks 19 and 20) or increase in Hgb by ≥ 1.2 g/dL (average of Weeks 19 and 20) over pre-dose average (average of the two Hgb values obtained prior to dosing) without receiving ESA or transfusion. Participants were assigned to 1 of 3 study groups based on their ESA status at the screening visit: Naïve, Previously Treated and Actively Treated. Analysis of this secondary outcome measure was performed in the ESA Treatment Naïve group, defined as participants who had never received treatment with an ESA and who had a screening Hgb level of ≤10.5 g/dL.
Time Frame: Weeks 19 and 20
Population: MITT Population. Only participants with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 68 | 38
Percentage of participants | 50 | 7.9

5. Secondary Outcome: Percentage of Participants Achieving a Successful Hemoglobin Response in ESA Previously Treated Group
Description: Hgb response was defined as participants with mean Hgb ≥11.0 g/dL (average of Weeks 19 and 20) or increase in Hgb by ≥ 1.2 g/dL (average of Weeks 19 and 20) over pre-dose average (average of the two Hgb values obtained prior to dosing) without receiving ESA or transfusion. Participants were assigned to 1 of 3 study groups based on their ESA status at the screening visit: Naïve, Previously Treated and Actively Treated. Analysis of this secondary outcome measure was performed in the ESA Previously Treated group, defined as participants who had previously received ≥1 dose of an ESA, had been off of ESA therapy for ≥11 weeks at the time of screening, and had a screening Hgb level of ≤10.5 g/dL.
Time Frame: Weeks 19 and 20
Population: MITT Population. Only participants with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 41 | 21
Percentage of participants | 41.5 | 19
Statistical Analysis 1: Comparison: Vadadustat vs Placebo; Test type: Other; p = 0.0953, Fisher Exact

6. Secondary Outcome: Percentage of Participants Achieving a Successful Hemoglobin Response in ESA Actively Treated Group
Description: Hgb response was defined as participants with mean Hgb ≥11.0 g/dL (average of Weeks 19 and 20) or increase in Hgb by ≥ 1.2 g/dL (average of Weeks 19 and 20) over pre-dose average (average of the two Hgb values obtained prior to dosing) without receiving ESA or transfusion. Participants were assigned to 1 of 3 study groups based on their ESA status at the screening visit: Naïve, Previously Treated and Actively Treated. Analysis of this secondary outcome measure was performed in the ESA Actively Treated group, defined as participants who had been actively treated with an ESA for a minimum of 4 months before screening, had received at least 2 doses within the last 4 months, had received their last dose within 6 weeks before screening, and had a screening Hgb level ≥9.5 g/dL and ≤12.0 g/dL.
Time Frame: Weeks 19 and 20
Population: MITT Population. Only participants with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 27 | 13
Percentage of participants | 33.3 | 7.7
Statistical Analysis 1: Comparison: Vadadustat vs Placebo; Test type: Other; p = 0.1238, Fisher Exact

7. Secondary Outcome: Percentage of Participants Achieving a Successful Hemoglobin Response, Analyzed in mITT Population
Description: Hgb response was defined as participants with mean Hgb ≥11.0 g/dL (average of Weeks 19 and 20) or increase in Hgb by ≥ 1.2 g/dL (average of Weeks 19 and 20) over pre-dose average (average of the two Hgb values obtained prior to dosing) without receiving ESA or transfusion. Analysis of this secondary outcome measure was performed in the mITT population.
Time Frame: Weeks 19 and 20
Population: MITT Population. Only participants with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 136 | 72
Percentage of participants | 44.1 | 11.1
Statistical Analysis 1: Comparison: Vadadustat vs Placebo; Test type: Other; p < 0.0001, Fisher Exact

8. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Blood samples were collected to assess Hgb. Baseline was defined as the mean of two samples obtained prior to dosing (Screening and Baseline). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. A positive change from Baseline indicated Hgb concentration increased.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 12, Week 16, Week 19 and Week 20
Population: MITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 135 | 72
g/dL
  Baseline | 9.94 (0.861) | 9.96 (0.790)
  Week 2: number analyzed (Participants) | 131 | 70
  Week 2 | 0.1 (0.756) | -0.22 (0.564)
  Week 4: number analyzed (Participants) | 126 | 68
  Week 4 | 0.39 (0.868) | -0.25 (0.679)
  Week 6: number analyzed (Participants) | 123 | 67
  Week 6 | 0.63 (1.059) | -0.41 (0.835)
  Week 8: number analyzed (Participants) | 124 | 67
  Week 8 | 0.69 (1.087) | -0.4 (0.878)
  Week 12: number analyzed (Participants) | 121 | 64
  Week 12 | 0.9 (1.066) | -0.2 (0.864)
  Week 16: number analyzed (Participants) | 113 | 64
  Week 16 | 0.76 (1.055) | -0.18 (0.963)
  Week 19: number analyzed (Participants) | 110 | 56
  Week 19 | 0.73 (1.063) | -0.16 (0.926)
  Week 20: number analyzed (Participants) | 105 | 63
  Week 20 | 0.88 (1.161) | -0.08 (0.933)
Statistical Analysis 1: Comparison: Vadadustat vs Placebo; Week 2; Test type: Other; p = 0.0019, t-test, 2 sided
Statistical Analysis 2: Comparison: Vadadustat vs Placebo; Week 4; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Vadadustat vs Placebo; Week 6; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Vadadustat vs Placebo; Week 8; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 5: Comparison: Vadadustat vs Placebo; Week 12; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 6: Comparison: Vadadustat vs Placebo; Week 16; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 7: Comparison: Vadadustat vs Placebo; Week 19; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 8: Comparison: Vadadustat vs Placebo; Week 20; Test type: Other; p < 0.0001, t-test, 2 sided

9. Secondary Outcome: Absolute Values of Hemoglobin
Description: Blood samples were collected at indicated time points for analysis of hemoglobin
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 12, Week 16, Week 19 and Week 20
Population: MITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 135 | 72
g/dL
  Baseline | 9.94 (0.861) | 9.96 (0.79)
  Week 2: number analyzed (Participants) | 132 | 70
  Week 2 | 10.02 (0.909) | 9.74 (0.714)
  Week 4: number analyzed (Participants) | 127 | 68
  Week 4 | 10.35 (0.979) | 9.7 (0.733)
  Week 6: number analyzed (Participants) | 123 | 67
  Week 6 | 10.61 (0.996) | 9.6 (0.758)
  Week 8: number analyzed (Participants) | 124 | 67
  Week 8 | 10.66 (0.987) | 9.6 (0.848)
  Week 12: number analyzed (Participants) | 121 | 64
  Week 12 | 10.87 (0.958) | 9.82 (0.682)
  Week 16: number analyzed (Participants) | 113 | 64
  Week 16 | 10.79 (0.895) | 9.83 (0.841)
  Week 19: number analyzed (Participants) | 110 | 56
  Week 19 | 10.74 (0.881) | 9.93 (0.897)
  Week 20: number analyzed (Participants) | 105 | 63
  Week 20 | 10.88 (1.002) | 9.93 (0.859)

10. Secondary Outcome: Change From Baseline in Hematocrit
Description: Blood samples were collected to assess Hematocrit. Baseline was defined as the mean of two samples obtained prior to dosing (Screening and Baseline). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. A positive change from Baseline indicated Hematocrit concentration increased.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 12, Week 16, Week 19 and Week 20
Population: MITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 135 | 72
Percentage of red blood cells in blood
  Baseline | 30.4 (2.96) | 30.3 (2.90)
  Week 2: number analyzed (Participants) | 132 | 70
  Week 2 | 0.8 (2.46) | -0.6 (1.97)
  Week 4: number analyzed (Participants) | 127 | 68
  Week 4 | 2 (2.87) | -0.5 (2.33)
  Week 6: number analyzed (Participants) | 122 | 67
  Week 6 | 2.5 (3.55) | -1 (2.87)
  Week 8: number analyzed (Participants) | 124 | 67
  Week 8 | 2.7 (3.44) | -1 (3.15)
  Week 12: number analyzed (Participants) | 121 | 64
  Week 12 | 3 (3.5) | -0.3 (2.95)
  Week 16: number analyzed (Participants) | 113 | 64
  Week 16 | 3.3 (3.48) | -0.1 (3.24)
  Week 19: number analyzed (Participants) | 110 | 56
  Week 19 | 3.1 (3.51) | 0 (3.19)
  Week 20: number analyzed (Participants) | 105 | 63
  Week 20 | 3 (3.8) | 0.1 (3.13)
Statistical Analysis 1: Comparison: Vadadustat vs Placebo; Week 2; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Vadadustat vs Placebo; Week 4; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Vadadustat vs Placebo; Week 6; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Vadadustat vs Placebo; Week 8; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 5: Comparison: Vadadustat vs Placebo; Week 12; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 6: Comparison: Vadadustat vs Placebo; Week 16; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 7: Comparison: Vadadustat vs Placebo; Week 19; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 8: Comparison: Vadadustat vs Placebo; Week 20; Test type: Other; p < 0.0001, t-test, 2 sided

11. Secondary Outcome: Absolute Values of Hematocrit
Description: Blood samples were collected at indicated time points for analysis of Hematocrit.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 12, Week 16, Week 19 and Week 20
Population: MITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 135 | 72
Percentage of red blood cells in blood
  Baseline | 30.4 (2.96) | 30.3 (2.9)
  Week 2: number analyzed (Participants) | 132 | 70
  Week 2 | 31.2 (3.06) | 29.7 (2.62)
  Week 4: number analyzed (Participants) | 127 | 68
  Week 4 | 32.4 (3.17) | 29.7 (2.72)
  Week 6: number analyzed (Participants) | 122 | 67
  Week 6 | 33.1 (3.21) | 29.4 (2.46)
  Week 8: number analyzed (Participants) | 124 | 67
  Week 8 | 33.2 (3.05) | 29.3 (3.05)
  Week 12: number analyzed (Participants) | 121 | 64
  Week 12 | 33.5 (3.19) | 30.2 (2.05)
  Week 16: number analyzed (Participants) | 113 | 64
  Week 16 | 34 (3.02) | 30.3 (2.87)
  Week 19: number analyzed (Participants) | 110 | 56
  Week 19 | 33.7 (2.83) | 30.7 (2.83)
  Week 20: number analyzed (Participants) | 105 | 63
  Week 20 | 33.6 (3.19) | 30.4 (2.7)

12. Secondary Outcome: Change From Baseline in Red Blood Cell Count
Description: Blood samples were collected to assess red blood cell count. Baseline was defined as the mean of two samples obtained prior to dosing (Screening and Baseline). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. A positive change from Baseline indicated red blood cell count increased.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 12, Week 16, Week 19 and Week 20
Population: MITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 10^6 cells per microliter
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 135 | 72
10^6 cells per microliter
  Baseline | 3.38 (0.402) | 3.34 (0.322)
  Week 2: number analyzed (Participants) | 132 | 70
  Week 2 | 0.02 (0.243) | -0.08 (0.212)
  Week 4: number analyzed (Participants) | 127 | 68
  Week 4 | 0.12 (0.277) | -0.08 (0.222)
  Week 6: number analyzed (Participants) | 123 | 67
  Week 6 | 0.18 (0.346) | -0.14 (0.276)
  Week 8: number analyzed (Participants) | 124 | 67
  Week 8 | 0.23 (0.351) | -0.14 (0.32)
  Week 12: number analyzed (Participants) | 121 | 64
  Week 12 | 0.3 (0.357) | -0.08 (0.29)
  Week 16: number analyzed (Participants) | 113 | 64
  Week 16 | 0.28 (0.363) | -0.06 (0.331)
  Week 19: number analyzed (Participants) | 110 | 56
  Week 19 | 0.26 (0.374) | -0.04 (0.319)
  Week 20: number analyzed (Participants) | 105 | 63
  Week 20 | 0.3 (0.411) | -0.01 (0.314)
Statistical Analysis 1: Comparison: Vadadustat vs Placebo; Week 2; Test type: Other; p = 0.0031, t-test, 2 sided
Statistical Analysis 2: Comparison: Vadadustat vs Placebo; Week 4; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Vadadustat vs Placebo; Week 6; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Vadadustat vs Placebo; Week 8; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 5: Comparison: Vadadustat vs Placebo; Week 12; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 6: Comparison: Vadadustat vs Placebo; Week 16; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 7: Comparison: Vadadustat vs Placebo; Week 19; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 8: Comparison: Vadadustat vs Placebo; Week 20; Test type: Other; p < 0.0001, t-test, 2 sided

13. Secondary Outcome: Absolute Values of Red Blood Cell Count
Description: Blood samples were collected at indicated time points for analysis of red blood cell count.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 12, Week 16, Week 19 and Week 20
Population: MITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 10^6 cells per microliter
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 135 | 72
10^6 cells per microliter
  Baseline | 3.38 (0.402) | 3.34 (0.322)
  Week 2: number analyzed (Participants) | 132 | 70
  Week 2 | 3.39 (0.418) | 3.25 (0.321)
  Week 4: number analyzed (Participants) | 127 | 68
  Week 4 | 3.51 (0.409) | 3.24 (0.317)
  Week 6: number analyzed (Participants) | 123 | 67
  Week 6 | 3.57 (0.412) | 3.2 (0.321)
  Week 8: number analyzed (Participants) | 124 | 67
  Week 8 | 3.61 (0.421) | 3.21 (0.377)
  Week 12: number analyzed (Participants) | 121 | 64
  Week 12 | 3.68 (0.457) | 3.27 (0.295)
  Week 16: number analyzed (Participants) | 113 | 64
  Week 16 | 3.69 (0.44) | 3.29 (0.343)
  Week 19: number analyzed (Participants) | 110 | 56
  Week 19 | 3.67 (0.415) | 3.32 (0.332)
  Week 20: number analyzed (Participants) | 105 | 63
  Week 20 | 3.7 (0.453) | 3.33 (0.318)

14. Secondary Outcome: Change From Baseline in Reticulocyte Count
Description: Blood samples were collected to assess reticulocyte count. Baseline was defined as mean of two samples obtained prior to dosing (Screening and Baseline). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. A positive change from Baseline indicated reticulocyte count increased.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 12, Week 16, Week 19 and Week 20
Population: MITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 10^6 cells per microliter
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 136 | 72
10^6 cells per microliter
  Baseline: number analyzed (Participants) | 136 | 71
  Baseline | 2.12 (0.858) | 1.97 (0.816)
  Week 2: number analyzed (Participants) | 128 | 68
  Week 2 | 0.61 (0.778) | -0.07 (0.532)
  Week 4: number analyzed (Participants) | 126 | 66
  Week 4 | 0.29 (0.686) | 0.06 (0.485)
  Week 6: number analyzed (Participants) | 121 | 66
  Week 6 | 0.19 (0.749) | 0.08 (0.549)
  Week 8: number analyzed (Participants) | 124 | 64
  Week 8 | -0.08 (0.737) | 0.06 (0.665)
  Week 12: number analyzed (Participants) | 121 | 63
  Week 12 | -0.12 (0.742) | 0.02 (0.639)
  Week 16: number analyzed (Participants) | 110 | 61
  Week 16 | 0.03 (0.678) | -0.03 (0.659)
  Week 19: number analyzed (Participants) | 108 | 55
  Week 19 | 0.07 (0.88) | -0.05 (0.672)
  Week 20: number analyzed (Participants) | 105 | 61
  Week 20 | 0.03 (0.666) | 0.12 (0.786)
Statistical Analysis 1: Comparison: Vadadustat vs Placebo; Week 2; Test type: Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Vadadustat vs Placebo; Week 4; Test type: Other; p = 0.0133, t-test, 2 sided
Statistical Analysis 3: Comparison: Vadadustat vs Placebo; Week 6; Test type: Other; p = 0.3053, t-test, 2 sided
Statistical Analysis 4: Comparison: Vadadustat vs Placebo; Week 8; Test type: Other; p = 0.1918, t-test, 2 sided
Statistical Analysis 5: Comparison: Vadadustat vs Placebo; Week 12; Test type: Other; p = 0.2090, t-test, 2 sided
Statistical Analysis 6: Comparison: Vadadustat vs Placebo; Week 16; Test type: Other; p = 0.6184, t-test, 2 sided
Statistical Analysis 7: Comparison: Vadadustat vs Placebo; Week 19; Test type: Other; p = 0.3604, t-test, 2 sided
Statistical Analysis 8: Comparison: Vadadustat vs Placebo; Week 20; Test type: Other; p = 0.4056, t-test, 2 sided

15. Secondary Outcome: Absolute Values of Reticulocyte Count
Description: Blood samples were collected at indicated time points for analysis of reticulocyte count.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 12, Week 16, Week 19 and Week 20
Population: MITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 10^6 cells per microliter
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 136 | 72
10^6 cells per microliter
  Baseline: number analyzed (Participants) | 136 | 71
  Baseline | 2.12 (0.858) | 1.97 (0.816)
  Week 2: number analyzed (Participants) | 128 | 68
  Week 2 | 2.74 (1.069) | 1.91 (0.727)
  Week 4: number analyzed (Participants) | 126 | 66
  Week 4 | 2.44 (0.962) | 2.06 (0.731)
  Week 6: number analyzed (Participants) | 121 | 66
  Week 6 | 2.32 (0.996) | 2.07 (0.897)
  Week 8: number analyzed (Participants) | 124 | 64
  Week 8 | 2.05 (0.884) | 2.09 (0.85)
  Week 12: number analyzed (Participants) | 121 | 63
  Week 12 | 2.02 (0.959) | 2 (0.846)
  Week 16: number analyzed (Participants) | 110 | 61
  Week 16 | 2.13 (0.992) | 1.96 (0.83)
  Week 19: number analyzed (Participants) | 108 | 56
  Week 19 | 2.21 (1.297) | 1.92 (0.77)
  Week 20: number analyzed (Participants) | 105 | 61
  Week 20 | 2.17 (0.954) | 2.1 (0.88)

16. Secondary Outcome: Percentage of Participants Who Received ESA Rescue
Description: Participants were administered epoetin alfa or darbepoetin alfa as a rescue medication who met the Hgb rescue criteria in addition to having experienced a clinically significant worsening of their anemia or the symptoms of anemia.
Time Frame: Up to 20 Weeks
Population: MITT Population. Only participants with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 136 | 72
Percentage of participants
  Epoetin Alfa | 4.4 | 12.5
  Darbepoetin Alfa | 0 | 4.2

17. Secondary Outcome: Mean Number of ESA Rescue Doses Administered Per Participant
Description: Participants were administered epoetin alfa or darbepoetin alfa as a rescue medication who have met the Hgb rescue criteria in addition to having experienced a clinically significant worsening of their anemia or the symptoms of anemia.
Time Frame: Up to 20 Weeks
Population: MITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Doses/participants
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 6 | 9
Doses/participants
  Epoetin Alfa | 1.7 (1.63) | 2.8 (1.79)
  Darbepoetin Alfa: number analyzed (Participants) | 0 | 3
  Darbepoetin Alfa |  | 4.3 (2.52)

18. Secondary Outcome: Percentage of Participants Who Received Packed Red Blood Cell Transfusion Rescue
Description: Participants were administered packed red blood cell transfusion as a rescue medication who have met the Hgb rescue criteria in addition to having experienced a clinically significant worsening of their anemia or the symptoms of anemia
Time Frame: Up to 20 Weeks
Population: MITT Population. Only participants with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 136 | 72
Percentage of participants | 0 | 1.4

19. Secondary Outcome: Number of Packed Red Blood Cell Transfusion Administered Per Participant
Description: Participants were administered packed red blood cells as a rescue medication who have met the Hgb rescue criteria in addition to having experienced a clinically significant worsening of their anemia or the symptoms of anemia.
Time Frame: Up to 20 Weeks
Population: MITT Population. Only participants who received transfusion rescue were analyzed.
Measure: Median (Full Range); unit: Units of blood per participant
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 0 | 1
Units of blood per participant |  | 1.0 [1 to 1]

20. Secondary Outcome: Time to First Transfusion or ESA Rescue Medication Intake
Description: Rescue therapy was defined as red blood cell transfusion or ESA administration in participants meeting Hgb rescue criteria in addition to having experienced a clinically significant worsening of their anemia or the symptoms of anemia.
Time Frame: Up to 20 Weeks
Population: MITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 136 | 72
Weeks | 21.6 (6.08) | 21.2 (5.71)
Statistical Analysis 1: Comparison: Vadadustat vs Placebo; Test type: Other; p = 0.0017, Log Rank; Hazard Ratio (HR) = 4.1451, 95% CI 2-sided [1.5752 to 10.9080]

21. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence, signs, symptoms, disease, or laboratory or physiological observations occurring in a participant administered with drug, regardless of a causal relationship with that treatment or usage. This also included all suspected adverse medication reactions, reactions from medication overdose, abuse, withdrawal, sensitivity, toxicity, unrelated illnesses, including worsening a pre-existing condition, injury, or accidents. Serious Adverse Events (SAEs) was defined as any life-threatening condition; hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; or death.
Time Frame: Up to 20 Weeks
Population: Intent-to-treat (ITT) population included all randomized participants who received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 138 | 72
Participants
  TEAEs | 58 | 29
  Treatment-emergent SAEs | 33 | 11

22. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Parameter Values
Description: Parameters assessed for laboratory values included hematology, serum chemistry, and urinalysis. The investigator was responsible for reviewing laboratory results for clinically significant changes.
Time Frame: Up to 20 Weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 138 | 72
Participants
  Hematology | 0 | 0
  Serum chemistry | 1 | 0
  Urinalysis | 0 | 0

23. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Parameters assessed for vital signs included sitting (at rest for a minimum of 5 minutes) heart rate, respiratory rate, body temperature, and blood pressure. The investigator was responsible for reviewing laboratory results for clinically significant changes.
Time Frame: Up to 20 Weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 138 | 72
Participants | 0 | 0

24. Secondary Outcome: Number of Participants With Clinically Abnormal 12-Lead Electrocardiogram (ECG) Findings
Description: A standard 12-lead ECG was performed following dosing in a supine position for approximately 10 minutes. ECGs were taken prior to blood draws when possible. The investigator was responsible for reviewing laboratory results for clinical significance.
Time Frame: Up to 20 Weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 138 | 72
Participants | 1 | 0

25. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Physical Examination Findings
Description: A Baseline physical examination was performed at screening. Otherwise, abbreviated physical examinations were conducted and were to include heart, lung, and abdomen. The investigator was responsible for reviewing laboratory results for clinically significant changes.
Time Frame: Up to 20 Weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 138 | 72
Participants | 0 | 0

26. Other Pre Specified Outcome: Exploratory: Change From Baseline in Iron and Total Iron Binding Capacity (TIBC)
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Exploratory: Change From Baseline in Transferrin
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Exploratory: Change From Baseline in Transferrin Saturation
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Exploratory: Mean Weekly Dose of Intravenous Elemental Iron Administered
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Exploratory: Absolute Values of Iron and Total Iron Binding Capacity (TIBC)
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Exploratory: Absolute Values of Transferrin
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Exploratory: Absolute Values of Transferrin Saturation
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Exploratory: Absolute Values of Reticulocyte Hemoglobin Content
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Exploratory: Change From Baseline in Reticulocyte Hemoglobin Content
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Exploratory: Change From Baseline in Hemoglobin A1c
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Exploratory: Absolute Values of Hemoglobin A1c
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Exploratory: Absolute Values of Lipids
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Exploratory: Change From Baseline in Lipids
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Exploratory: Change From Baseline in Hepcidin
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

40. Other Pre Specified Outcome: Exploratory: Absolute Values of Hepcidin
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

41. Other Pre Specified Outcome: Exploratory: Change From Baseline in Vascular Endothelial Growth Factor (VEGF)
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

42. Other Pre Specified Outcome: Exploratory: Absolute Values of Interleukin 6, Cystatin C, Intact Parathyroid Hormone, and Calcitonin
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

43. Other Pre Specified Outcome: Exploratory: Change From Baseline in Interleukin 6, Cystatin C, Intact Parathyroid Hormone, and Calcitonin
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

44. Other Pre Specified Outcome: Exploratory: Neurocognitive Functioning as a Measure
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

45. Other Pre Specified Outcome: Exploratory: Patient-Reported Outcome Measures
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

46. Other Pre Specified Outcome: Exploratory: Plasma Concentrations of Vadadustat and Its Glucuronide Metabolites
Time Frame: Baseline and up to Week 20
Reporting Status: Not Posted

47. Other Pre Specified Outcome: Exploratory: Plasma Concentrations of Vadadustat and Its Glucuronide Metabolites
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the start of treatment (Day 1) up to 24 weeks.
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events (AEs) that began (or pre-existing AEs that worsened) on or after the first dose through each participant's last participation date, were reported.
Arm/Group | Vadadustat | Placebo
All-Cause Mortality (participants affected / at risk) | 3/138 | 0/72
Serious Adverse Events (participants affected / at risk) | 33/138 | 11/72
Other Adverse Events (participants affected / at risk) | 58/138 | 29/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vadadustat (N=138) | Placebo (N=72)
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 1 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
ASTHENIA (General disorders) | 1 | 0
FATIGUE (General disorders) | 1 | 0
SUDDEN CARDIAC DEATH (General disorders) | 1 | 0
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 | 0
ANGIOEDEMA (Immune system disorders) | 1 | 0
CELLULITIS (Infections and infestations) | 1 | 0
CRYPTOSPORIDIOSIS INFECTION (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 1
OSTEOMYELITIS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 2 | 1
PNEUMONIA INFLUENZAL (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
UROSEPSIS (Infections and infestations) | 0 | 1
CEREBRAL HAEMORRHAGE TRAUMATIC (Injury, poisoning and procedural complications) | 1 | 0
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 | 0
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 2 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
DIABETIC AUTONOMIC NEUROPATHY (Nervous system disorders) | 1 | 0
HYPOGLYCAEMIC UNCONSCIOUSNESS (Nervous system disorders) | 1 | 0
PRESYNCOPE (Nervous system disorders) | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 1
DIABETIC NEPHROPATHY (Renal and urinary disorders) | 1 | 0
GOODPASTURE'S SYNDROME (Renal and urinary disorders) | 1 | 0
KIDNEY FIBROSIS (Renal and urinary disorders) | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 7 | 2
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 6 | 0
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 1 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACCELERATED HYPERTENSION (Vascular disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 1 | 0
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vadadustat (N=138) | Placebo (N=72)
Diarrhoea (Gastrointestinal disorders) | 14 | 3
Nausea (Gastrointestinal disorders) | 14 | 3
Constipation (Gastrointestinal disorders) | 5 | 4
Fatigue (General disorders) | 11 | 5
Oedema peripheral (General disorders) | 10 | 7
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 5
Urinary tract infection (Infections and infestations) | 8 | 6
Headache (Nervous system disorders) | 8 | 2
Dizziness (Nervous system disorders) | 7 | 3
Hypertension (Vascular disorders) | 11 | 2
Hypotension (Vascular disorders) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other